CLINICAL TRIAL: NCT05502263
Title: Interest of Maximal Oxygen Uptake and Ventilatory Inefficiency (VE/VCO2 Slope) Measured During Cardiopulmonary Exercise Test on Morbidity and Mortality of Lung Resection Candidates
Brief Title: Interest of CPET to Predict Mortality and Complications of Lung Resection Candidates
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Université Libre de Bruxelles (Other)
Responsible Party: Principal Investigator, Kevin Forton, PhD, Université Libre de Bruxelles
Other Study IDs: 2021293
Record Dates: First submitted 2022-08-12; First posted 2022-08-16 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Exercise Test; Thoracic Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- moderate/high risk: FEV and/or DLCO <80% And VO2peak <20ml/kg.min or <75% predicted value
- Control: FEV and DLCO >80% and VO2peak > 20ml/kg.min or >75% predicted value

SUMMARY:
Anatomic lung resection is the treatment of choice for the management of cancerous lung nodules Non-Small-Cell Lung Carcinoma (NSCLC). Systematic functional evaluation can reduce the risk of mortality and morbidity of candidates. Scientific societies recommend a cardiac and spirometry evaluation (including pulmonary diffusion capacity). In this context, patients with FEV1 or less than 80% of the predicted value are subjected to a more thorough evaluation of the physical physical capacity by cardiopulmonary exercise test (CPET) to determine VO2 max (Brunelli et al 2009). Patients with a VO2 max <35% of predicted values or <10ml/kg/min, or a postoperative predicted value of DLCO or FEV1(ppoDLCO, ppoVEMS) less than 30% associated with a postoperative VO2max less than 35% or 10 ml/min/kg should be offered an alternative treatment option (Begum et al 2016). In contrast, a VO2max greater than 20ml/min/kg is considered at low surgical risk (Brunelli et al 2009).

For patients with a VO2 max between 10 and 20ml/kg/min, operability depends on the extent of the resection. In this group of patients, other parameters measured with CPET could be used to optimize the selection of patients given the inability of some the inability of some patients to provide a maximal effort, thus resulting in a sub-maximal evaluation of physical capacity.

The VE/VCO2 slope, ventilatory equivalents or chronotropic recovery are parameters classically used in classically used in heart failure and have recently been shown to be independent prognostic factors as independent prognostic factors for 90-day and 2-year mortality after anatomical lung resection. Moreover, these factors do not depend on the maximality of the test and could again help us to risk-stratify for a sub-maximal and therefore not optimal test.

ELIGIBILITY:
Inclusion Criteria: Lobectomy or Segmentectomy or Wedge Resection for Non-Small Cell Lung cancer

- Performed CPET

Exclusion Criteria:

* pulmonary resection for diagnostic
* pneumonectomies and any extensive resections (chest wall-associated resections, Pancoast tumors, resection of the atrium or superior vena cava, resection of the diaphragm, spinal resection, pleuro-pneumonectomy, tracheal sleeve pneumonectomy, intrapericardial pneumonectomy), as well as metastases, benign lesions, and any other non-oncologic pulmonary resections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lobectomy or Segmentectomy or Wedge Resection for a patient Non-Small Cell Lung cancer patient
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Mortality | within 30 days after surgery
  death
Mortality | within 12 months after surgery
  death
Major respiratory complication in hospital | within 30 days after surgery
  pneumonia (chest roentgenogram infiltrates/consolidation, leukocytosis, fever)
  * respiratory failure needng mechanical ventilation for longer than 48 hours, adult respiratory distress syndrome
Minor respiratory complication in hospital | within 30 days after surgery
  air leak >5 day (Patient experienced a postoperative air leak for >5 days),atelectasis requiring bronchoscopy, atrial or ventricular arrhythmia, Empyema, Wound infection, delirium, renal failure

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Forton, PhD, Principal Investigator — Erasme University Hospital ULB
Locations (1):
- Erasme Hospital, Brussels, Belgium

REFERENCES:
- [Background] Brunelli A, Belardinelli R, Pompili C, Xiume F, Refai M, Salati M, Sabbatini A. Minute ventilation-to-carbon dioxide output (VE/VCO2) slope is the strongest predictor of respiratory complications and death after pulmonary resection. Ann Thorac Surg. 2012 Jun;93(6):1802-6. doi: 10.1016/j.athoracsur.2012.03.022. Epub 2012 May 4. PMID 22560968